CLINICAL TRIAL: NCT05228483
Title: Safety and Efficacy of Carbon Dioxide（CO2）Fractional Laser Combined With Photodynamic Therapy in the Treatment of Female Vulvar Lichen Sclerosus
Brief Title: Carbon Dioxide（CO2）Fractional Laser Plus Photodynamic Therapy in Female Patients With Vulvar Lichen Sclerosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XijingH-PF-20211102
Record Dates: First submitted 2021-12-22; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-11

CONDITIONS: Vulva Lichen Sclerosus
Keywords: vulva lichen sclerosus; female; CO2 Fractional Laser; Photodynamic Therapy
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Aminolevulinic Acid; Mometasone Furoate; Ointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodynamic treatment monotherapy or combined with CO2 fractional laser (Experimental): For patients who receive photodynamic therapy, lesions will be symmetrically randomized into two sides. One side will receive 5-aminolevulinic acid (5-ALA) with a red light illumination(80mW/cm2, and 120J/ cm2); while the other side will receive CO2 fractional laser(parameter: 20mm *20mm, spot coverage rate 10%, and 18-25mJ/cm2) before photodynamic therapy. Treating area should cover 0.5cm beyond the visible boundary of the lesion. In total 6 therapies will be given for each patient, with 14±3d intervals.
  Interventions: Device: CO2 fractional laser; Combination Product: 5-aminolevulinic acid (5-ALA) with red light illumination
- Mometasone furoate cream (Active Comparator): Mometasone furoate cream (0.1%) for topical application, frequency: once daily, 5 days/week, for the first month; once every other day, for the second month; twice a week for the third month; the area of application should cover 0.5cm beyond the visible boundary of the lesion.
  Interventions: Drug: Mometasone furoate (MMF) 0.1% ointment

INTERVENTIONS:
Device: CO2 fractional laser — CO2 fraction laser
  Arms: Photodynamic treatment monotherapy or combined with CO2 fractional laser
Combination Product: 5-aminolevulinic acid (5-ALA) with red light illumination — 5-aminolevulinic acid (5-ALA) is a photosensitizing agent which can induce photochemical reactions in tissues in response to an appropriate wavelength of light (red light 630-635nm).
  Arms: Photodynamic treatment monotherapy or combined with CO2 fractional laser
Drug: Mometasone furoate (MMF) 0.1% ointment — 0.1% Mometasone furoate ointment is a potent steroid and has been proven to result as efficacious and well tolerated as clobetasol propionate which represent the recomended first-line treatment of vulvar lichen sclerosus.
  Arms: Mometasone furoate cream

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of CO2 fractional laser combined with photodynamic therapy in female patients with vulvar lichen sclerosus.

DETAILED DESCRIPTION:
This is a randomized, open-labeled, assessor-blind, parallel control study. 134 enrolled patients will be randomized to apply either topical 0.1% corticosteroid mometasone furoate(MMF) ointment or photodynamic therapy.

For patients who receive photodynamic therapy, lesions will be symmetrically randomized into two sides. One side will receive CO2 fractional laser before photodynamic therapy, while the other side will receive photodynamic therapy only.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 (inclusive), female patients;
2. present typical clinical manifestations of of vulvar lichen sclerosus, confirmed by histopathological examination;
3. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Severe organic diseases, such as severe heart, lung, liver, kidney insufficiency, coagulation dysfunction, etc.;
2. Suffer from autoimmune diseases, such as systemic lupus erythematosus, thyroid disease, etc.;
3. Suffer from photoallergic diseases, such as chronic photosensitivity dermatitis, plant solar dermatitis;
4. People with porphyria or porphyria allergy;
5. Suffer from psychiatric diseases, such as schizophrenia, etc.;
6. Those who are undergoing systemic treatment due to malignant tumor diseases, such as cervical cancer;
7. It is confirmed by laboratory pathogenic screening to have syphilis, HIV, and other sexually transmitted diseases or viral hepatitis;
8. Patients with current bacterial or fungal infections in the anus and genitals;
9. Women of childbearing age who have pregnancy plans, are pregnant, or are breastfeeding during the observation period of this study;
10. Patients who are systematically using glucocorticoids, immunosuppressants, and anticoagulants;
11. Use glucocorticoids for topical or local injection and calcineurin inhibitors for topical use within 4 weeks;
12. Those who are allergic to 5-aminolevulinic acid or its base, mometasone furoate or its base;
13. Other situations that the investigator considers inappropriate to participate in the clinical study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Global Subjective Score 75（GSS75） rate | 2 weeks after the final treatment
  GSS75 is defined as ≥75% improvement from baseline in global subjective score using pain and itching visual analog scales with score from 0 (absent) to 10 (most severe imaginable). GSS75 rate is the rate of patients achieving GSS75.

SECONDARY OUTCOMES:
Recurrence rate | 6 months, 12 months after the final treatment
  Recurrence rate: the number of patients relapse/the number of patients who completed all treatment. Relapse is defined as an increase of 1 point in any of the six indicators of GOS, or an increase of ≥ 3 points in any of the GSS, or an increase of 1 point in any of the QOL compared with that at the 2-week visit after the final treatment.
Global Subjective Score 75（GSS75） | 12 weeks after the final treatment
  GSS75 is defined as ≥75% improvement from baseline in global subjective score using pain and itching visual analog scales with score from 0 (absent) to 10 (most severe imaginable)
Global Objective Score（GOS） | 2 weeks, 12 weeks, 6 months, 12 months after the final treatment
  Sum of scores in 6 aspects: Erythema, leukoplakia, hyperkeratosis, purpuric lesions, degree of sclerosis, scar-like atrophy (0 = absent, 1 = mild, 2 = moderate, 3 = severe). Range : 0 - 18.
Lichen Sclerosus Area （LSA） | 2 weeks, 12 weeks, 6 months, 12months after the final treatment
  The improvement of lichen sclerosus area from baseline by photograph documents with a standard scale
Quality of Life（QOL） | 2 weeks, 12 weeks, 6 months, 12 months after the final treatment
  Sum of scores of four indexes: dysuria, defecation difficulty, dysesthesia and dyspareunia (applicable patients) ( 0 = absent, 1 = mild, 2 = moderate, 3 = severe). Range: 0-12.
Dermoscope Area Score （DAS） | 2 weeks, 12 weeks, 6 months, 12 months after the final treatment
  Dermoscope assessment of vessel morphology, bright white or white- yellowish structureless areas, shiny white streaks, purple dots, peppering blue-gray dots, erosions, and rose petal sign ( 0 = absent, 1 = mild, 2 = moderate, 3 = severe).
incidence of adverse events | up to 12 months
  incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Guannan Zhu, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No